CLINICAL TRIAL: NCT01089543
Title: A Multi-Center, Randomized, Double-Blind Study of E3810 for Japanese Subjects With Functional Dyspepsia
Brief Title: A Study of E3810 for Japanese Subjects With Functional Dyspepsia (SAMURAI Study: Suppression of Acid Milieu With Rabeprazole Improving Functional Dyspepsia ) (Study E3810-J081-204)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E3810-J081-204
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Results first posted 2013-11-19 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-11

CONDITIONS: Functional Dyspepsia
Keywords: dyspepsia; rabeprazole; Japan
MeSH Terms: conditions — Dyspepsia | interventions — Rabeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Rabeprazole 10 mg (Experimental)
  Interventions: Drug: Rabeprazole
- Rabeprazole 20 mg (Experimental)
  Interventions: Drug: Rabeprazole
- Rabeprazole 40 mg (Experimental)
  Interventions: Drug: Rabeprazole
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rabeprazole — Rabeprazole 10 mg tablet taken orally once daily after breakfast for 8 weeks.
  Other Names: E3810
  Arms: Rabeprazole 10 mg
Drug: Rabeprazole — Rabeprazole 20 mg tablet taken orally once daily after breakfast for 8 weeks.
  Other Names: E3810
  Arms: Rabeprazole 20 mg
Drug: Rabeprazole — Rabeprazole 40 mg tablet taken orally once daily after breakfast for 8 weeks.
  Other Names: E3810
  Arms: Rabeprazole 40 mg
Drug: Placebo — Rabeprazole Placebo tablet taken orally once daily after breakfast for 8 weeks.
  Other Names: E3810
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of rabeprazole compared to placebo in Japanese subjects with Functional Dyspepsia.

ELIGIBILITY:
Inclusion criteria:

-Participants diagnosed as Functional Dyspepsia according to Rome III criteria.

Exclusion criteria:

* Participants with neuropsychiatric disorder.
* Participants diagnosed with irritable bowel syndrome, inflammatory bowel disease and serious constipation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiumi Okubo, Study Director — Eisai Co., Ltd.
Locations (46):
- Japan (46):
  - Nagoya, Aichi-ken
  - Akita, Akita
  - Chikushino-shi, Fukuoka
  - Fukuoka, Fukuoka
  - Kitakyushu, Fukuoka
  - Gifu, Gifu
  - Maebashi, Gunma
  - Hiroshima, Hiroshima
  - Sapporo, Hokkaido
  - Kobe, Hyōgo
  - Nishinomiya, Hyōgo
  - Tsuchiura, Ibaraki
  - Takamatsu, Kagawa-ken
  - Kagoshima, Kagoshima-ken
  - Yokohama, Kanagawa
  - Kochi, Kochi
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Sendai, Miyagi
  - Miyazaki, Miyazaki
  - Ōita, Oita Prefecture
  - Yufu, Oita Prefecture
  - Nakagami, Okinawa
  - Hirakata, Osaka
  - Moriguchi, Osaka
  - Osaka, Osaka
  - Suita, Osaka
  - Takatsuki, Osaka
  - Karatsu, Saga-ken
  - Saga, Saga-ken
  - Saitama, Saitama
  - Kusatsu, Shiga
  - Izumo, Shimane
  - Fujieda, Shizuoka
  - Hamamatsu, Shizuoka
  - Shizuoka, Shizuoka
  - Ōtawara, Tochigi
  - Shimotsuga, Tochigi
  - Bunkyo, Tokyo
  - Mitaka, Tokyo
  - Nakano City, Tokyo
  - Ōta-ku, Tokyo
  - Setagaya City, Tokyo
  - Shibuya City, Tokyo
  - Shinagawa, Tokyo
  - Yamagata, Yamagata

REFERENCES:
- [Derived] Iwakiri R, Tominaga K, Furuta K, Inamori M, Furuta T, Masuyama H, Kanke K, Nagahara A, Haruma K, Kinoshita Y, Higuchi K, Takahashi S, Kusano M, Iwakiri K, Kato M, Hongo M, Hiraishi H, Watanabe S, Miwa H, Naito Y, Fujimoto K, Arakawa T. Randomised clinical trial: rabeprazole improves symptoms in patients with functional dyspepsia in Japan. Aliment Pharmacol Ther. 2013 Oct;38(7):729-40. doi: 10.1111/apt.12444. Epub 2013 Aug 20. PMID 23957383

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 66 centers in Japan during the period of 21-April-2010 to 12-Aug-2011.
Pre-assignment Details: Participants were initially enrolled into a 1- or 2-week run-in period (single-blinded administration of placebo). Participants who did not respond to placebo were randomized to an 8-week treatment period (double-blinded administration) of rabeprazole 10 mg, 20 mg, 40 mg, or placebo, once daily after breakfast.
Groups:
- Rabeprazole 10 mg: Rabeprazole 10 mg tablet taken orally once daily after breakfast for 8 weeks.
- Rabeprazole 20 mg: Rabeprazole 20 mg tablet taken orally once daily after breakfast for 8 weeks.
- Rabeprazole 40 mg: Rabeprazole 40 mg tablet taken orally once daily after breakfast for 8 weeks.
Period: Overall Study
Arm/Group | Rabeprazole 10 mg | Rabeprazole 20 mg | Rabeprazole 40 mg | Placebo
Started | 84 | 85 | 84 | 85
Completed | 81 | 81 | 81 | 83
Not Completed | 3 | 4 | 3 | 2
Not completed — Withdrawal by Subject | 2 | 3 | 3 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Per Protocol Set (PPS): was defined as those participants who complied with the study protocol. N= 338 participants were enrolled at study start. However, a total of 307 participants were included in PPS for efficacy evaluation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rabeprazole 10 mg | Rabeprazole 20 mg | Rabeprazole 40 mg | Placebo | Total
Number analyzed (Participants) | 77 | 76 | 74 | 80 | 307
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (14.9) | 50.2 (16.5) | 46.4 (14.8) | 45.8 (15.5) | 47.3 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 40 | 47 | 44 | 174
  Male | 34 | 36 | 27 | 36 | 133

OUTCOME MEASURES:

1. Primary Outcome: Rate of Complete Dyspepsia Symptom Relief
Description: The rate of complete dyspepsia symptom relief according to the Dyspepsia Symptom Questionnaire (DSQ) was defined as a score of 1 for all four major dyspeptic symptoms at week 8 and according to the diary defined as all four dyspepsia symptoms recorded absent during the 7 days prior to week 8. Values presented as percentage of participants.
Time Frame: Up to 8 Weeks (including 7 days prior)
Population: Per Protocol Set (PPS) population defined as those participants who complied with the study protocol.
Measure: Number; unit: Percentage of Participants
Arm/Group | Rabeprazole 10 mg | Rabeprazole 20 mg | Rabeprazole 40 mg | Placebo
Number analyzed (Participants) | 77 | 76 | 74 | 80
Percentage of Participants
  DSQ (n= 76, n= 75, n= 74, n= 78) | 22.4 | 29.3 | 27.0 | 17.9
  Diary Recordings (n= 77, n= 76, n=74, n=80) | 22.1 | 28.9 | 27.0 | 17.5

2. Secondary Outcome: Rate of Satisfactory Symptom Relief
Description: The rate of satisfactory symptom relief according to the DSQ defined as scores of <= 2 for all four major dyspepsia symptoms at week 8 and the diary recordings defined as a frequency of <= 1 day for all four major dyspepsia symptoms during the 7 days before week 8. Lastly, treatment success according to the participants' impression questionnaire where participants answered "yes" or "no" when asked if given the choice, whether they would want to continue to take the study drug after clinical trial completion. Values presented as percentage of participants.
Time Frame: Up to 8 Weeks (including 7 days prior)
Population: Per Protocol Set (PPS) Population: defined as those participants who complied with the study protocol.
Measure: Number; unit: Percentage of participants
Arm/Group | Rabeprazole 10 mg | Rabeprazole 20 mg | Rabeprazole 40 mg | Placebo
Number analyzed (Participants) | 77 | 76 | 74 | 80
Percentage of participants
  DSQ (n=76, n=75, n=74, n=78) | 42.1 | 45.3 | 39.2 | 28.2
  Diary Recordings (n=77, n=76, n=74, n=80) | 37.7 | 48.7 | 39.2 | 30.0
  Treatment Success (n=76, n=75, n=74, n=78) | 72.4 | 85.3 | 64.9 | 59.0

ADVERSE EVENTS:
Time Frame: Up to 8 weeks
Description: Safety Analysis Set was defined as those participants who received at least one dose of study drug (N= 338). One participant was incorrectly assigned to a different dose group.
Arm/Group | Rabeprazole 10 mg | Rabeprazole 20 mg | Rabeprazole 40 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/85 | 1/85 | 1/83 | 1/85
Other Adverse Events (participants affected / at risk) | 28/85 | 20/85 | 31/83 | 22/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rabeprazole 10 mg (N=85) | Rabeprazole 20 mg (N=85) | Rabeprazole 40 mg (N=83) | Placebo (N=85)
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rabeprazole 10 mg (N=85) | Rabeprazole 20 mg (N=85) | Rabeprazole 40 mg (N=83) | Placebo (N=85)
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 2 | 2
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Periodontitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 3 | 1
Gastroenteritis (Infections and infestations) | 0 | 3 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 10 | 7 | 15 | 4
Pharyngitis (Infections and infestations) | 0 | 1 | 1 | 3
Aspartate Aminotransferase Increased (Investigations) | 2 | 0 | 1 | 0
Blood Triglycerides Increased (Investigations) | 3 | 0 | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 4
Headache (Nervous system disorders) | 3 | 3 | 1 | 0
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No